CLINICAL TRIAL: NCT03708185
Title: Does Beta-alanine Supplementation Augment the Skeletal Muscle Adaptive Response to 8 Weeks of High-intensity Interval Training
Brief Title: Beta-alanine Supplementation and High-intensity Interval Training
Acronym: BEAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 180509/B/02
Record Dates: First submitted 2018-06-12; First posted 2018-10-17 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Healthy
MeSH Terms: interventions — beta-Alanine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Doubly-blinded & randomised using an online randomisation website.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT + beta-alanine (Experimental): Participants will ingest an active supplement containing beta-alanine for a period of 12 weeks. During the last 8 weeks of that period, participants will take part in a structured program of high-intensity interval training.
  Interventions: Dietary Supplement: Beta-alanine
- HIIT + placebo (Experimental): Participants will ingest a placebo supplement containing no beta-alanine for a period of 12 weeks. During the last 8 weeks of that period, participants will take part in a structured program of high-intensity interval training.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beta-alanine — N/A: see arm description
  Arms: HIIT + beta-alanine
Dietary Supplement: Placebo — N/A: see arm description
  Arms: HIIT + placebo

SUMMARY:
The present study will seek to quantify whether a period of HIIT alongside β-alanine supplementation will improve the adaptation to training, and therefore performance, more than a period of HIIT alone.

DETAILED DESCRIPTION:
Whilst high-intensity interval training (HIIT) is a powerful stimulus to increase endurance exercise performance, there are potential nutritional interventions that can be put in place to further increase performance gains.

Energy for the contraction of muscles is created in the mitochondria. HIIT can improve the function of mitochondria, therefore improving performance.

Β-alanine is a commonly used supplement that can improve exercise performance by increasing the amount of carnosine in muscle. Carnosine has many functions that may help improve exercise capacity.

The present study will seek to quantify whether a period of HIIT alongside β-alanine supplementation will improve the adaptation to training, and therefore performance, more than a period of HIIT alone.

ELIGIBILITY:
Inclusion Criteria:

* Moderately trained (vo2max: 50 - 60 ml/kg/min).
* Females must be taking an oral contraceptive, or using a contraceptive implant.

Exclusion Criteria:

* A recent history of musculoskeletal injury
* Diagnosed cardiovascular or metabolic disease
* Regular use of beta-alanine supplements

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline work done on a cycle ergometer in a cycling capacity test at 110%VO2max following a period of 4 weeks of beta-alanine supplementation and then 8 weeks of beta-alanine supplementation and high intensity interval training | At weeks 0, 4 and 12 of study.
  Subjects will have previously performed an incremental test to exhaustion (VO2max test). A work-load that corresponds to 110 % of the peak power output (Wmax) will be calculated, and participants will be asked to cycle at this power output until volitional exhaustion. This test will be preceded but a bout of 90-minute cycling at 65%VO2max. Tests will be performed on a Lode Excalibur Sport, and software linked to the bike will record data.

SECONDARY OUTCOMES:
VO2max | At weeks 0, 4, 8 and 12 of study.
  VO2max will be determined from data collected through a metabolic cart. It will be measured during an incremental test to exhaustion performed on a cycle ergometer.
Substrate utilisation | At weeks 0, 4 and 12 of study.
  Substrate utilisation will be calculated from data collected through a metabolic cart and its software. It will be measured during the 90-minute steady-state cycle for 4 periods of 3 minutes. Carbohydrate and lipid oxidation rates will be calculated using equations by Jeukendrup & Wallis (2005).
Muscle carnosine concentration | At weeks 0, 4 and 12 of study.
  Using the Bergstrom muscle biopsy technique. Samples will be frozen immediately in liquid nitrogen and will be later analysed using validated techniques
Muscle enzyme (citrate synthase, hexokinase, β-HAD, PFK) activity | At weeks 0, 4 and 12 of study.
  Using the Bergstrom muscle biopsy technique. Samples will be frozen immediately in liquid nitrogen and will be later analysed using validated techniques
Muscle buffering capacity | At weeks 0, 4 and 12 of study.
  Using the Bergstrom muscle biopsy technique. Samples will be frozen immediately in liquid nitrogen and will be later analysed using validated techniques
Muscle metabolites (AMP, ADP, ATP, Pi, IMP, PCr, Cr, lactate, pyruvate, NAD+/NADH, glucose, G6P, citrate) | At weeks 0, 4 and 12 of study.
  Using the Bergstrom muscle biopsy technique. Samples will be frozen immediately in liquid nitrogen and will be later analysed using validated techniques
Muscle gene expression | At weeks 0, 4 and 12 of study.
  Using the Bergstrom muscle biopsy technique. Samples will be frozen immediately in liquid nitrogen and will be later analysed using validated techniques
Plasma metabolites (NEFA, glucose, glycerol, lactate) | At weeks 0, 4 and 12 of study.
  A cannula will be used to draw blood from subjects at several time points. Whole blood will be centrifuged immediately and its plasma split into aliquots and stored in a -80°C freezer for later analysis.
Heart rate | At weeks 0, 4 and 12 of study, and through whole training period (weeks 8-12)
  Heart rate will be measured throughout with the use of a heart rate monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Davenport, MSc, Principal Investigator — The University of Exeter
Locations (1):
- School of Sport and Health Sciences, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No